CLINICAL TRIAL: NCT04616092
Title: Effect of Preoperative Intravenous Ferric Carboxymaltose on Postoperative Transfusion Reduction in Anemia Patients Scheduled for Clipping Surgery for Unruptured Intracranial Aneurysms
Brief Title: Effect of Preoperative Intravenous Ferric Carboxymaltose for Clipping Surgery
Acronym: PICASA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: Vifor Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SeoulNUBH_NS
Record Dates: First submitted 2020-10-26; First posted 2020-11-04 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-10

CONDITIONS: Cerebral Aneurysm Unruptured; Iron Deficiency Anemia; Surgery
MeSH Terms: conditions — Anemia, Iron-Deficiency

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- FERINJECT Group (Experimental): Patients with FERINJECT injection
  Interventions: Drug: FEFINJECT
- Observation Group (No Intervention): Patients without FERINJECT injection

INTERVENTIONS:
Drug: FEFINJECT — FEFINJECT injection
  Arms: FERINJECT Group

SUMMARY:
Hypothesis: Correction of preoperative anemia can reduce the need for intra-/postoperative RBC transfusions and can improve surgical outcomes.

DETAILED DESCRIPTION:
Anemia is one of the major risk factors that has been shown to compromise surgical outcome in many fields of surgery. Although red blood cell (RBC) transfusions can be used to correct anemia quickly, RBC transfusions are known to be a risk factor that worsens the outcome of surgery. In cerebrovascular disease, anemia can decrease the delivery of oxygen to brain tissue and can cause cerebral ischemia, which can lead to secondary brain damage. On the other hand, RBC transfusion may increase the viscosity of the blood, thereby reducing the cerebral blood flow, or causing side effects such as vasospasm or thromboembolic event. Therefore, there is a growing need for measures to correct anemia and reduce the number of transfusions in the treatment of cerebrovascular diseases.

The effectiveness of ferric carboxymaltose for postoperative anemia correction in orthopedic and general surgery has been reported in several studies. However, researches on the effect of ferric carboxymaltose to correct preoperative anemia is rare, and there has been no study on the efficacy of ferric carboxymaltose, especially in brain surgery. However, as the population of the elderly grows and the technology of inspection develops, the number of diagnosis of cerebrovascular diseases increases. In particular, the incidence of unruptured intracranial aneurysms (UIA) has increased by 29.7% every year since 2008. Accordingly, clipping sugery, known as the treatment of UIA, has increased by 16.0% every year since 2008.21 Therefore, it is necessary to study the efficacy of ferric carboxymaltose to correct the anemia and to decrease the number of transfusion in clipping surgery for UIA.

Seicean et al. analyzed the effects of preoperative anemia and RBC transfusion on the surgical outcomes of 668 patients who underwent surgery for intracranial aneurysms for 7 years. 29.6 % of 668 patients were diagnosed with anemia, preoperatively. 28.3 % of patients with anemia, and 8.1 % of patients without anemia received RBC transfusions, intra-/postoperatively. Patients with preoperative anemia showed significantly higher frequency of RBC transfusions (p<0.01) in general cohort, and hospital length of stay (LOS) (p<0.01) and the rate of major complications (p=0.02) was significantly higher in the group receiving RBC transfusions. This study have reported that preoperative anemia was predictive of perioperative transfusion in the general and matched cohorts (data not shown). Other studies also demostrated that lower preoperative hemoglobin was assodiated with perioperative transfusion.

Investigators performed 427 patients who underwent clipping surgery for UIAs in 2017 in single institute (Seoul National University Bundang Hospital), where has the biggest cerebrovascular center in Korea and is one of the world's best hospitals for cerebrovascular surgery. Among 427 patients, Investigators retrospectively analysed the relationship between preoperative anemia and postoperative transfusion for 338 patients treated for UIA sized under 15mm and located in anterior circulation to maintain patient consistency. 15.4% of patients who underwent clipping surgery were diagnosed with anemia before surgery. Though Investigators did not check the level of ferritin or transferrin saturation, most patients were suspected of IDA because all patients had no chronic inflammatory disease or underlying disease causing anemia. The mean amount of intraoperative bleeding was 484.5ml, and 45.7% of the patients were given intra-/postoperative transfusion. In conclusion, the frequency of intra-/postoperative RBC transfusion was significantly higher in patients diagnosed with preoperative anemia. (p<0.01) Based on these results, investigators hypothesized that correcting anemia before surgery could reduce the need for postoperative RBC transfusion and conducted a pilot study. From November 2018 to April 2019, FERINJECT 500mg was administered to 12 patients who underwent clipping surgery for UIAs. The average haemoglobin (Hb) increased from 11.4g/dl before FERINJECT to 13.1g/dl on the day of surgery. Three patients (25.0%) received a transfusion after surgery. When investigators retrospectively compared the group with patients without correcting the anemia, investigators concluded that the anemia corrected group significantly lowered the probability of postoperative transfusion. (p <0.01) Accordingly, investigators designed a prospective study to evaluate the effect of preoperative anemia correction using FERINJECT on the need for RBC transfusion and surgical outcome in patients undergoing clipping surgery for UIAs.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients: 19≤ age < 80
2. Patients with IDA (All of the following conditions must be met) A. Hb: female (10≤Hb<12g/dl), male (10≤Hb<13g/dl) B. Ferritin < 100ng/ml C. Transferrin saturation<20%
3. Patients with UIAs A. UIAs located in anterior circulation B. Size < 15mm C. Operable with clipping alone

Exclusion Criteria:

1. Age: <19, ≥80
2. Hb<10
3. Anemia except IDA A. Anaplastic anemia B. Hemolytic anemia C. Anemia with chronic disease
4. UIAs located in posterior circulation
5. Size of UIA ≥ 15mm
6. Not operable with clipping alone

Ages: 19 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2020-11 (Estimated); Primary Completion 2022-11 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Red Blood Cell transfusion rate in packs | 7 days after operation
  Reduction of transfusion rate per patient in hospital resulting from administration of intravenous ferric carboxymaltose for the patients who undergoing clipping surgery

SECONDARY OUTCOMES:
Anemia correction (Hemoglobin in g/dl) | 1 day before sugery
  Effect of preoperative intravenous ferric carboxymaltose administration on anemia correction in patients with anemia before clipping surgery
Adverse event rate and hospital length of stay (LOS) in days | Within 30days after operation
  Effect of preoperative intravenous ferric carboxymaltose administration on reduction of adverse event and hospital LOS after clipping surgery

CONTACTS AND LOCATIONS:
Overall Officials: Si Un Lee, Professor, Principal Investigator — Seoul National University Bundang Hospital

IPD SHARING:
Plan to Share IPD: No
If requested by the publisher, a serial number can be assigned and shared.

REFERENCES:
- [Background] Dhar R, Zazulia AR, Videen TO, Zipfel GJ, Derdeyn CP, Diringer MN. Red blood cell transfusion increases cerebral oxygen delivery in anemic patients with subarachnoid hemorrhage. Stroke. 2009 Sep;40(9):3039-44. doi: 10.1161/STROKEAHA.109.556159. Epub 2009 Jul 23. PMID 19628806
- [Background] Hendrickson JE, Hillyer CD. Noninfectious serious hazards of transfusion. Anesth Analg. 2009 Mar;108(3):759-69. doi: 10.1213/ane.0b013e3181930a6e. PMID 19224780
- [Background] Rosenberg NF, Koht A, Naidech AM. Anemia and transfusion after aneurysmal subarachnoid hemorrhage. J Neurosurg Anesthesiol. 2013 Jan;25(1):66-74. doi: 10.1097/ANA.0b013e31826cfc1d. PMID 23047622
- [Background] Oddo M, Milby A, Chen I, Frangos S, MacMurtrie E, Maloney-Wilensky E, Stiefel M, Kofke WA, Levine JM, Le Roux PD. Hemoglobin concentration and cerebral metabolism in patients with aneurysmal subarachnoid hemorrhage. Stroke. 2009 Apr;40(4):1275-81. doi: 10.1161/STROKEAHA.108.527911. Epub 2009 Mar 5. PMID 19265059
- [Background] Naidech AM, Shaibani A, Garg RK, Duran IM, Liebling SM, Bassin SL, Bendok BR, Bernstein RA, Batjer HH, Alberts MJ. Prospective, randomized trial of higher goal hemoglobin after subarachnoid hemorrhage. Neurocrit Care. 2010 Dec;13(3):313-20. doi: 10.1007/s12028-010-9424-4. PMID 20717750
- [Background] Naidech AM, Jovanovic B, Wartenberg KE, Parra A, Ostapkovich N, Connolly ES, Mayer SA, Commichau C. Higher hemoglobin is associated with improved outcome after subarachnoid hemorrhage. Crit Care Med. 2007 Oct;35(10):2383-9. doi: 10.1097/01.CCM.0000284516.17580.2C. PMID 17717494
- [Result] Beattie WS, Karkouti K, Wijeysundera DN, Tait G. Risk associated with preoperative anemia in noncardiac surgery: a single-center cohort study. Anesthesiology. 2009 Mar;110(3):574-81. doi: 10.1097/ALN.0b013e31819878d3. PMID 19212255
- [Result] Dunne JR, Malone D, Tracy JK, Gannon C, Napolitano LM. Perioperative anemia: an independent risk factor for infection, mortality, and resource utilization in surgery. J Surg Res. 2002 Feb;102(2):237-44. doi: 10.1006/jsre.2001.6330. PMID 11796024
- [Result] Kulier A, Levin J, Moser R, Rumpold-Seitlinger G, Tudor IC, Snyder-Ramos SA, Moehnle P, Mangano DT; Investigators of the Multicenter Study of Perioperative Ischemia Research Group; Ischemia Research and Education Foundation. Impact of preoperative anemia on outcome in patients undergoing coronary artery bypass graft surgery. Circulation. 2007 Jul 31;116(5):471-9. doi: 10.1161/CIRCULATIONAHA.106.653501. Epub 2007 Jul 9. PMID 17620512
- [Result] Musallam KM, Tamim HM, Richards T, Spahn DR, Rosendaal FR, Habbal A, Khreiss M, Dahdaleh FS, Khavandi K, Sfeir PM, Soweid A, Hoballah JJ, Taher AT, Jamali FR. Preoperative anaemia and postoperative outcomes in non-cardiac surgery: a retrospective cohort study. Lancet. 2011 Oct 15;378(9800):1396-407. doi: 10.1016/S0140-6736(11)61381-0. Epub 2011 Oct 5. PMID 21982521
- [Derived] Lee SU, Sung SB, Koo CH, Lim S, Lee SH, Choi TW, Kim YD, Ban SP, Kwon OK, Bang JS. Effect of Preoperative Intravenous Ferric Carboxymaltose on Postoperative Transfusion Reduction in Iron Deficiency Anemia Patients Scheduled for Clipping Surgery for Unruptured Intracranial Aneurysms: The PICASA Trial - A Single Center, Single-Blind Randomized Clinical Trial. Anaesth Crit Care Pain Med. 2025 Oct 24;45(2):101646. doi: 10.1016/j.accpm.2025.101646. Online ahead of print. PMID 41342691